CLINICAL TRIAL: NCT03986749
Title: Biological Augmentation With Subacromial Bursa in Arthroscopic Rotator Cuff Repair - Postoperative Findings Using Doppler Ultrasonography
Brief Title: Bursa Augmentation in Arthroscopic Rotator Cuff Repair
Acronym: ARCR-Bursa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: OE-0116 (ARCR-BursaSeries)
Record Dates: First submitted 2019-06-05; First posted 2019-06-14 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Rotator Cuff Tear or Rupture, Not Specified as Traumatic
Keywords: arthroscopic rotator cuff repair; bursa augmentation; neovascularization; Doppler ultrasonography
MeSH Terms: conditions — Rotator Cuff Injuries; Rupture; Neovascularization, Pathologic

STUDY DESIGN:
Intervention Model Description: prospective observational case-series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARCR-BursaSeries (Experimental): Tendon healing in the reconstruction of the rotator cuff, taking advantage of augmentation potential of the subacromial bursa.
  Interventions: Procedure: Doppler ultrasonography after bursa augmentation

INTERVENTIONS:
Procedure: Doppler ultrasonography after bursa augmentation — Dynamic ultrasound examination with Grading of blood vessels using the modified Ohberg Score in the longitudinal scan in dynamic ultrasound of the rotator cuff tendon - primary to surgery and 3 weeks later.

SUMMARY:
The aim of this first study is to investigate in a case series through sequential sonographic imaging, using Doppler ultrasonography, the postoperative morphology, especially vascularity and findings of neovascularity, after bursa augmentation in arthroscopic rotator cuff repair.

DETAILED DESCRIPTION:
The outcome of rotator cuff (RC) reconstruction with and without bursa augmentation, considering also the inflammatory status of the bursa, will be systematically investigated for the first time. The influencing role of the inflammatory status of the bursa, of the RC tendon and the synovial membrane at the time of the operation on the tendinous healing rate, the patient-relevant outcome factors and the revision rate will be assessed. In a further approach, basic knowledge about the role of bursa inflammation and its influence in the development and regeneration of tendon pathologies shall be gained. The findings of the whole project could lead to improve tendon healing in the reconstruction of the rotator cuff, taking advantage of augmentation potential of the subacromial bursa.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and older
* Patient with C-shaped posterosuperior rotator cuff tear (SSP / ± ISP, ± SCP Tear Lafosse ≤ 1 (SCP no repair, only debridement))
* Retraction ≤ 2 according to Patte
* Fatty infiltration ≤ 2 according to Goutallier
* Eligible for arthroscopic double row rotator cuff repair in Suture Bridge technique.
* Written informed consent

Exclusion Criteria:

* Legal incompetence
* Last subacromial cortisone infiltration ≤ 6 months
* Systemic rheumatologic-inflammatory disease
* Diabetes Mellitus
* Smoker

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Dynamic ultrasound examination with grading of blood vessels | 3 months
  using the modified Ohberg Score

SECONDARY OUTCOMES:
Tendon integrity | 6 months
  intact / partially ruptured / ruptured
Tendon condition | 6 months
  Thickness of the repaired tendons (mm)
Range of motion | 6 months
  Elevation (flexion), abduction, external rotation by 0° abduction, external-internal rotation by 90° abduction
Shoulder muscle strength | 6 months
  Shoulder strength in 90° Abduction (kg) measured using a spring balance
Oxford Shoulder Score (OSS) | 6 months
  Patient-reported Oxford Shoulder Score from 0 (worse) to 48 (best)
Subjective shoulder value (SSV) | 6 months
  Patient-reported Subjective shoulder value from 0 (worse) to 100% (best)
Constant Murley score (CMS) | 6 months
  Constant Murley functional score from 0 (worse) to 100 (best)
Level of satisfaction | 6 months
  Level of satisfaction using Number Rating Scale from 0 (not satisfied) to 10 (highly satisfied)
EQ-5D utilities | 6 months
  Patient-reported Quality of life (EuroQol EQ-5D-5L) as Utility index from 0 (worse) to 1 (best health)
Adverse events | 6 months
  Number of patients with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Markus Scheibel, MD, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No